CLINICAL TRIAL: NCT00881491
Title: Treatment Outcome With a Revascularization Protocol Using the Triple Versus Double Antibiotic Paste
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Kenneth Hargreaves, Chair, Department of Endodontics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20090181H
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Pulp Necrosis
Keywords: Regeneration (revascularization) of dental pulp; Immature permanent tooth with a diagnosis of
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Group A - Double antibiotic paste: intracanal medicament consisting of ciprofloxacin and metronidazole
  Interventions: Drug: Double Antibiotic Paste
- Group B (Experimental): Group B - Triple Antibiotic Paste: intracanal medicament consisting of ciprofloxacin, metronidazole, minocycline
  Interventions: Drug: Triple Antibiotic Paste
- Group C (Active Comparator): Group C - Mineral trioxide aggregate: used as an apical barrier
  Interventions: Drug: Mineral Trioxide Aggregate

INTERVENTIONS:
Drug: Double Antibiotic Paste — ciprofloxacin and metronidazole powder mixed at a 1:1 ratio used as a intracanal medicament for disinfection.
  Arms: Group A
Drug: Triple Antibiotic Paste — ciprofloxacin, metronidazole & minocycline mixed to a 1:1:1 powder used as a intracanal medicament for disinfection.
  Arms: Group B
Drug: Mineral Trioxide Aggregate — standard material providing an apical barrier
  Arms: Group C

SUMMARY:
The purpose of this study is to determine the treatment outcomes in permanent teeth with necrotic pulp and immature root development that undergo a regenerative procedure using a triple antibiotic paste (ciprofloxacin, metronidazole, minocycline) versus a double antibiotic paste (ciprofloxacin, metronidazole)compared to the commonly used mineral trioxide aggregate (MTA) apexification treatment.

DETAILED DESCRIPTION:
Recent case series have reported positive outcomes treating necrotic immature permanent teeth with a regenerative procedure using a triple antibiotic paste (ciprofloxacin, metronidazole, minocycline). However, this method can result in considerable staining due to minocycline. In this randomized clinical trial, we will compare clinical outcomes of a triple antibiotic paste versus a double antibiotic paste (ciprofloxacin, metronidazole) intracanal medicament as compared to a standard treatment (immediate apexification with MTA) in permanent teeth with necrotic pulps and immature root development. We hypothesize there will be no significant differences between radiographic measures of root development after treatment with either the double versus triple antibiotic paste, and that both methods will produce significantly greater increases in root length and width compared to standard treatment. The primary outcome measures will be radiographic measurement of root length and dentinal wall thickness and the secondary outcomes will be lack of clinical symptoms and crown staining.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of pulpal necrosis with apical periodontitis
* patients 7-60 years of age
* maxillary or mandibular restorable single rooted immature permanent tooth with open apices
* acceptance of treatment plan with revascularization procedure
* healthy patient (ASA Class I or II physical status) with no systemic health problems

Exclusion Criteria:

* non-restorable teeth
* patients with ASA Class III or IV physical status (Immuno-compromised patients including patients who self-report to be a carrier of HIV, undergoing steroid therapy, or those who self-report with genetic or systemic diseases that could result in reduced immune response.
* child subjects unable to give assent

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures will be radiographic measurement of root length and dentinal wall thickness. | 3 measurements over 6 months
  1. st radiograph taken at 1 month post-procedure completion
  2. nd radiograph taken at 3 month post-procedure completion
  3. rd radiograph taken at 6 month post-procedure completion

SECONDARY OUTCOMES:
The secondary outcomes will be lack of clinical symptoms and crown staining. | assessed over the 6 month study period
  1. st clinical assessment done at 1 month post-procedure completion
  2. nd clinical assessment done at 3 month post-procedure completion
  3. rd clinical assessment done at 6 month post-procedure completion

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Hargreaves, DDS, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No data to be shared